CLINICAL TRIAL: NCT00601614
Title: Phase I Study of ZD6474 and Temozolomide in Patients With Advanced Cancer
Brief Title: Vandetanib and Temozolomide in Treating Patients With Advanced Solid Tumors That Cannot Be Removed By Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MC0615; MAYO-MC0615; MC0615; MAYO-07-004966
Record Dates: First submitted 2008-01-24; First posted 2008-01-28 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Temozolomide; vandetanib; Immunoenzyme Techniques

INTERVENTIONS:
Drug: temozolomide
Drug: vandetanib
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vandetanib together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vandetanib and temozolomide in treating patients with advanced solid tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of concurrently administered vandetanib and temozolomide in patients with unresectable, advanced solid tumors.
* To describe the toxicity profile of this regimen in these patients.
* To describe the response rate in patients treated with this regimen.
* To describe the effects of therapy on angiogenesis-related translational endpoints.

OUTLINE: Patients receive escalating doses of oral vandetanib once daily on days 1-28 and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and prior to each treatment course for correlative laboratory studies, including evaluation of plasma VEGF levels by ELISA, serum angiogenesis assay, and measurement of circulating endothelial cell populations (CD133, CD34, CD146). Frozen serum and plasma samples are also stored for future research studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor

  * Unresectable, advanced disease
* Measurable or evaluable disease
* No known standard therapy that is potentially curative or definitely capable of extending life expectancy exists
* No intracranial metastatic disease, unless it has been radiologically and clinically stable for the past 3 months

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/μL
* Absolute lymphocyte count > 1,000/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3 times ULN (≤ 5 times ULN if liver involvement)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance > 50 mL/min
* Potassium normal
* Serum calcium (ionized or adjusted for albumin) normal
* Magnesium normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No currently active diarrhea that results in an ongoing need for IV fluids and/or that may affect the ability of the patient to absorb vandetanib or tolerate diarrhea
* No evidence of severe or uncontrolled systemic disease or any concurrent condition that, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or that would jeopardize compliance with the study
* No other malignancies within the past 5 years, except cervical carcinoma in situ or adequately treated basal cell or squamous cell carcinoma of the skin
* No clinically significant cardiac event, such as myocardial infarction, NYHA class II-IV heart disease within the past 3 months, or presence of cardiac disease that, in the opinion of the treating physician, increases the risk of ventricular arrhythmia
* No history of arrhythmia (i.e., multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) that is symptomatic or requires treatment (CTCAE grade 3)

  * Atrial fibrillation that is controlled on medication allowed
* No asymptomatic sustained ventricular tachycardia
* No history of QTc prolongation as a result of other medication that required discontinuation of that medication
* No congenital long QT syndrome
* No 1st degree relative with unexplained sudden death under 40 years of age
* No left bundle branch block
* No QTc with Bazett's correction that is unmeasurable
* QTc < 480 msec on screening ECG
* No hypertension that is uncontrolled by medical therapy (i.e., systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg)
* No bleeding diathesis (inherited coagulopathy)

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 30 days since prior investigational agents
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin C or nitrosoureas)
* More than 4 weeks since prior immunotherapy or biologic therapy
* More than 4 weeks since prior major surgery

  * Surgical incision must be completely healed
* More than 4 weeks since prior radiotherapy, except palliative radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* No prior temozolomide or dacarbazine
* No prior enrollment in this study
* More than 2 weeks since prior and no concurrent known potent CYP3A4 inducers, such as rifampin, phenytoin, carbamazepine, barbiturates, or St. John's wort
* More than 2 weeks since prior and no concurrent drugs associated with an increased risk of causing Torsades de Pointes
* No concurrent medication that may cause QTc prolongation
* No concurrent anticoagulants
* No other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of vandetanib and temozolomide
Adverse events profile
Toxicity profile
Response profile
Time until any treatment-related toxicity
Time until treatment-related grade 3+ toxicity
Time until hematologic nadirs
Time to progression
Time to treatment failure
Correlation of changes in VEGF levels, serum angiogenesis, and circulating endothelial cells with response and dose levels

CONTACTS AND LOCATIONS:
Overall Officials: Ravi D. Rao, MD, MBBS, Study Chair — Mayo Clinic; Svetomir Markovic, MD, PhD — Mayo Clinic